CLINICAL TRIAL: NCT05998928
Title: A Clinical Study to Evaluate the Safety and Efficacy of BCMA-GPRC5D CAR-T in Patients With R/R MM Who Received Three or More Lines of Therapy
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of BCMA-GPRC5D CAR-T in Patients With Relapsed/Refractory Multiple Myeloma Who Received Three or More Lines of Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCMA-GPRC5D CAR-T-cells
Record Dates: First submitted 2023-07-28; First posted 2023-08-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + BCMA-GPRC5D CAR-T Cells (Experimental): Patients will receive lymphodepletion chemotherapy with fludarabine (30 mg/m2 body surface area) plus cyclophosphamide (300 mg/m2 body surface area) for 3 consecutive days during D-7 to D-3, followed by the infusion of BCMA-GPRC5D CAR-T cells at a single dose of 4.0×10^6/kg ± 50%/kg for one day.
  Interventions: Drug: Fludarabine + Cyclophosphamide + BCMA-GPRC5D CAR-T Cells

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + BCMA-GPRC5D CAR-T Cells — fludarabine 30 mg/m2 and cyclophosphamide 300 mg/m2 both on three consecutive days during D-7 to D-3
  BCMA-GPRC5D CAR-T Cells on day 0

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of bispecific BCMA-GPRC5D Chimeric antigen receptor (CAR) T-cells in patients with relapsed or refractory multiple myeloma who received three or more lines of therapy.

DETAILED DESCRIPTION:
B-cell maturation antigen (BCMA)-targeted Chimeric antigen receptor (CAR) T-cell therapy has yielded satisfactory clinical outcomes in patients with relapsed or refractory (R/R) multiple myeloma (MM). However, BCMA-targeted CAR-T cells cannot achieve a favorable response in patients with dim or negative BCMA expression on the tumor surface at baseline or relapse. G protein-coupled receptor, class C, group 5, member D (GPRC5D) is highly distributed on MM cells and proves to be a promising target for MM. In normal tissues, it is restrictedly expressed in hair follicle, rendering it a safe target for CAR-T cell therapy as well. To construct a bispecific BCMA-GPRC5D CAR structure would help mitigate the antigen escape and elevates the clinical efficacy.

This is an investigational study. The objectives are to evaluate the safety and efficacy of BCMA-GPRC5D CAR-T cells in adult patients with relapsed or refractory MM disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form;
2. Aged ≥ 18 years and ≤ 75 years;
3. Diagnosed as Multiple Myeloma (MM) according to the international standard for multiple myeloma (IMWG);
4. The presence of measurable disease at screening meets one of the following criteria:Serum M-protein ≥ 1.0 g/dL or Urine M-protein ≥ 200 mg/24h or diagnosed as Light-chain MM without measurable disease in serum and urine; Serum free light chain ≥ 10 mg/dL with an abnormal κ/λ ratio;
5. Patients must relapse or be refractory after three or more lines of therapy, which at least include: one Proteasome Inhibitor (PI), one Immunomodulatory Drug (IMiD), and one anti-CD38 monoclonal antibody;
6. diagnosed as relapsed/refractory disease or primary refractory disease;
7. The last treatment is ineffective, or the disease progresses within 60 days after the end of the last therapy;
8. Patients must recover from the toxicity of the last therapy (< grade 2 by CTCAE criteria);
9. ECOG score 1-2 points and the expected survival period ≥ 3 months;
10. Liver, kidney and cardiopulmonary functions meet the following requirements:

    1. Total bilirubin ≤ 1.5×ULN, alanine aminotransferase (ALT) ≤ 3 × ULN and aspartate aminotransferase (AST) ≤ 3 × ULN;
    2. Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 60 mL/min;
    3. Hemoglobin (Hb) ≥ 50 g/L without prior blood transfusion within 7 days;
    4. Baseline peripheral oxygen saturation > 92%;
    5. Corrected serum calcium ≤ 12.5 mg/dL (≤ 3.1 mmol/L) or free (ionized, ionic) calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L);
    6. Left ventricular ejection fraction (LVEF) > 45%, without confirmed pericardiac effusion and abnormal electrocardiography with clinical significance;
    7. Without clinically significant pleural effusion;
11. Venous access could be established; without contraindications of apheresis.

Exclusion Criteria:

1. Previous diagnosis and treatment of other malignancies within 3 years;
2. Patients received previous anti-tumor therapies before apheresis including following therapies: targeted therapies, epigenetics modulation drugs, other drugs or medical devices (invasive) of clinical trials, monoclonal antibodies, cytotoxic agents, PIs, IMiDs, radiotherapy;
3. Central Nervous System (CNS) involvement;
4. Patients with Fahrenheit macroglobulinemia, POEMS syndrome, or primary AL, amyloidosis;
5. Subjects with positive HBsAg or HBcAb positive and peripheral blood HBV DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive; HIV antibody positive; CMV DNA titer is higher than the lower limit of detection of the research institution; EBV DNA titer is higher than the lower limit of detection of the research institution;
6. Patients have a severe allergic history;
7. Patiens have severe systemic diseases or poor cardiovascular, liver, kidney functions;
8. Acute or chronic graft versus host disease (GvHD) occurs within 6 months before the screening or needs be treated with immunosuppressive agents;
9. Active autoimmune or inflammatory diseases of the nervous system;
10. Patients develop oncology emergencies and need to be treated before screening or infusion;
11. Uncontrolled infections that need antibiotics treatment;
12. Exposure to hematopoietic growth factor of cells within 1-2 weeks before apheresis;
13. Exposure to Corticosteriods or immunosuppressive agents within 2 weeks before apheresis;
14. Patients receive a major surgical operation within 4 weeks before lymphodepletion or do not recover completely before the enrollment; or plan to receive a major surgical operation during the study period;
15. Live attenuated vaccine within 4 weeks before screening;
16. Patients with severe mental illness;
17. Patients are addcited to alcohol or drugs;
18. Pregnant or Lactating Women; Patients and his or her spouse have a fertility plan within two years after CAR-T cell infusion;
19. Other conditions considered inappropriate by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome are graded by American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics - Cmax | within 2 years after infusion
  Cmax will be assessed from CAR T cell infusion to death or last follow-up (censored).
Pharmacokinetics and pharmacodynamics - Tmax | within 2 years after infusion
  Tmax will be assessed from CAR T cell infusion to death or last follow-up (censored).
Pharmacokinetics and pharmacodynamics - AUC 0-28d | within 2 years after infusion
  AUC 0-28d will be assessed from CAR T cell infusion to death or last follow-up (censored).
Pharmacokinetics and pharmacodynamics - AUC 0-90d | within 2 years after infusion
  AUC 0-90d will be assessed from CAR T cell infusion to death or last follow-up (censored).
Pharmacokinetics and pharmacodynamics - AUC 0-inf | within 2 years after infusion
  AUC 0-inf will be assessed from CAR T cell infusion to death or last follow-up (censored).
Pharmacokinetics and pharmacodynamics - AUC 0-t1/2 | within 2 years after infusion
  AUC 0-t1/2 will be assessed from CAR T cell infusion to death or last follow-up (censored).
Clinical efficacy of administering BCMA-GPRC5D CAR-T cells in Relapsed/Refractory multiple myeloma | within 2 years after infusion
  The rates of stringent complete response (sCRs), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR) will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall response rate (ORR) of administering BCMA-GPRC5D CAR-T cells in Relapsed/Refractory multiple myeloma. | within 2 years after infusion
  ORR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Clinical benefit rate | within 2 years after infusion
  Clinical benefit rate refers to ORR plus MR rate.
Duration of Response (DoR) of administering BCMA-GPRC5D CAR-T cells in Relapsed/Refractory multiple myeloma. | within 2 years after infusion
  DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Progress-free survival (PFS) of administering BCMA-GPRC5D CAR-T cells in Relapsed/Refractory multiple myeloma. | within 2 years after infusion
  PFS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival (OS) of administering BCMA-GPRC5D CAR-T cells in Relapsed/Refractory multiple myeloma. | within 2 years after infusion
  OS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Minimal Residual Disease (MRD) | within 2 years after infusion
  MRD status will be continuously monitored to assess the negative rate of MRD.
Antigen expression in tumor cells at different time points | within 2 years after infusion
  Changes in proportion of antigen-positive tumor cells after CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mailankody S, Devlin SM, Landa J, Nath K, Diamonte C, Carstens EJ, Russo D, Auclair R, Fitzgerald L, Cadzin B, Wang X, Sikder D, Senechal B, Bermudez VP, Purdon TJ, Hosszu K, McAvoy DP, Farzana T, Mead E, Wilcox JA, Santomasso BD, Shah GL, Shah UA, Korde N, Lesokhin A, Tan CR, Hultcrantz M, Hassoun H, Roshal M, Sen F, Dogan A, Landgren O, Giralt SA, Park JH, Usmani SZ, Riviere I, Brentjens RJ, Smith EL. GPRC5D-Targeted CAR T Cells for Myeloma. N Engl J Med. 2022 Sep 29;387(13):1196-1206. doi: 10.1056/NEJMoa2209900. PMID 36170501
- [Background] Fernandez de Larrea C, Staehr M, Lopez AV, Ng KY, Chen Y, Godfrey WD, Purdon TJ, Ponomarev V, Wendel HG, Brentjens RJ, Smith EL. Defining an Optimal Dual-Targeted CAR T-cell Therapy Approach Simultaneously Targeting BCMA and GPRC5D to Prevent BCMA Escape-Driven Relapse in Multiple Myeloma. Blood Cancer Discov. 2020 Sep;1(2):146-154. doi: 10.1158/2643-3230.BCD-20-0020. PMID 33089218